CLINICAL TRIAL: NCT01541345
Title: A Phase III, Randomized, Controlled Clinical Trial of Lateral Ridge Augmentation Using Autogenous Bone Blocks or Xenogenic Bone Block Grafts Loaded With Recombinant Human Bone Morphogenic Protein 2
Brief Title: Lateral Ridge Augmentation Using Autogenous Bone Blocks or Xenogenic Bone Block Grafts Loaded With Recombinant Human Bone Morphogenic Protein 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012DR2009
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (A) (Active Comparator): Bone augmentation will be performed using autogenous bone from the retromolar or chin area followed by a fixation with titanium screws at the recipients site; filled with deproteinized bovine bone mineral (DBBM) particles (Bio-Oss®, Geistlich Pharma AG, Wolhusen, Switzerland) and covered with a collagen membrane (Bio-Gide®, Geistlich Pharma AG, Switzerland). These course of action is well documented in the literature and standard procedures.
  Interventions: Device: Autogenous bone graft
- Test group (B) (Experimental): The bone augmentation will be performed using a deproteinized bovine bone mineral (DBBM) block (Bio-Oss Spongiosa Block®, Geistlich Parma AG, Wolhusen, Switzerland) and a collagen membrane (Bio-Gide®, Geistlich Pharma AG, Switzerland) similarly to the control group. In addition, DBBM will be loaded with rhBMPH-2 (InductOs®, Pfizer AG, Zurich, Switzerland).
  Interventions: Drug: InductOs; Procedure: Augmentation surgery

INTERVENTIONS:
Device: Autogenous bone graft — Bone augmentation will be performed using autogenous bone from the retromolar or chin area followed by a fixation with titanium screws at the recipients site; filled with deproteinized bovine bone mineral (DBBM) particles (Bio-Oss®, Geistlich Pharma AG, Wolhusen, Switzerland) and covered with a collagen membrane (Bio-Gide®, Geistlich Pharma AG, Switzerland)
  Arms: Control Group (A)
Drug: InductOs — CE-marked medical device Bio-Oss Spongiosa Block® (xenogenic bone) loaded with InductOs® (1.5 mg Dibotermin alfa / ml) covered with Bio-Gide® (collagen membrane). One time application at augmentation surgery.
  Arms: Test group (B)
Procedure: Augmentation surgery — CE-marked medical device Bio-Oss Spongiosa Block® (xenogenic bone) loaded with InductOs® (1.5 mg Dibotermin alfa / ml) covered with Bio-Gide® (collagen membrane)
  Arms: Test group (B)

SUMMARY:
Since there are no clinical studies available comparing the gold standard (autogenous bone graft plus resorbable membrane) to the promising combination of xenogenic bone graft loaded with rhBMP-2 in combination with a collagen membrane for localized ridge augmentation, the present exploratory study has been designed.

The aim of the present study is therefore to test whether or not the application of a xenogenic bone block loaded with rhBMP-2 will results in clinically, radiographically and histologically similar outcomes as the gold standard (autogenous bone block) for the regeneration of chronic ridge defects.

The investigators expect that there is no difference in bone quantity and quality between the two methods and that the use of the test treatment will be more user and patient friendly according to the patient perception/acceptance since no second surgical site will be necessary as well as cause less complications.

ELIGIBILITY:
Inclusion Criteria:

* requiring implant therapy for the reconstruction of 1 to 4 missing teeth
* revealing insufficient bone volume for implant placement (cases where less than 50% of the implant surface would be surrounded by native bone) requiring bone augmentation procedure

Exclusion Criteria:

* Medication with a contraindication for implant therapy
* Previous administration of InductOs
* Skeletal immaturity
* Any active malignancy or patient undergoing treatment for a malignancy
* An active infection at the operative site
* Persistent compartment syndrome or neurovascular residua of compartment syndrome
* Pathological fractures such as those observed in (but not limited to) Paget's disease or in metastatic bone
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Contraindications on ethical grounds,
* Pregnancy,
* Intention to become pregnant during the course of the study,
* Breast feeding,
* Treatment with other investigational products,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Patients where autogenous bone cannot be harvested.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04-25 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Bone quality/quantity | 4 month after augmentation surgery
  Bone quantity at 4 months after augmentation surgery, measured manually by ridge measurements and volumetrically on the basis of optical impressions and radiological assessment (X-ray and cone beam CT). Bone quality at 4 months after augmentation surgery, measured by histological assessment (yields different proportion per patient).

SECONDARY OUTCOMES:
Complications | 8 days and 4 month after augmentation surgery
  Complications (soft tissue, sensitivity) measured at suture removal (8 days after augmentation surgery) and 4 months after augmentation surgery. Any adverse events will be recorded for the treatment period from visit 1 to 4.
Bone quantity | at screening, augmentation surgery, suture removal, and during follow-up
  Bone quantity measured at screening, augmentation surgery, suture removal, and during follow-up
Patient's perception/acceptance | 8 days after augmentation surgery
  Patient's perception/acceptance (visual analogue scale VAS) measured at suture removal (8 days after augmentation surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Thoma, Prof. Dr., Principal Investigator — Clinic of Reconstructive Dentistry
Locations (2):
- Department of Oral Surgery & Radiology, Dental School, Medical University of Graz, Graz, Austria
- Center of Dental Medicine Clinic of Reconstructive Dentistry, Zurich, Switzerland